CLINICAL TRIAL: NCT01200680
Title: Genetic Clues to Chordoma Etiology: A Protocol to Identify Sporadic Chordoma Patients for Studies of Cancer-Susceptibility Genes
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910188; 10-C-N188
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-11-25

CONDITIONS: Genes; Sporadic Chordoma
Keywords: Pediatric and Adult; Gene Identification; Rare Bone Cancer; All Chordoma Sites; Natural History

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chordoma cohort: Chordoma patients

SUMMARY:
Background:

Chordoma is a rare, slow growing, often fatal bone cancer derived from remnants of the embryonic notochord. It occurs mostly in the axial skeleton (skull base, vertebrae, sacrum and coccyx), is more frequent in males than females, and has a median age at diagnosis of 58.5 years, with a wide age range. This typically sporadic tumor is often advanced at presentation, and mortality is high due to local recurrence or distant metastases. The usual treatment is surgery, followed by adjuvant radiation therapy. Chemotherapy has not had a significant treatment role. Reports of a small number of families worldwide with two or more relatives with chordoma support a role for susceptibility genes in chordoma etiology. Recently we determined that duplications of the T gene co-segregated with disease in four multiplex chordoma families. The T gene encodes brachyury, a tissue-specific transcription factor that is expressed in notochord cells and is essential for formation and maintenance of the notochord. Some of the other chordoma families that we studied did not have T-gene duplications; the aggregation of chordomas in these families may result from changes in other susceptibility genes or other types of mutations targeting the T gene. We are continuing gene identification studies of multiplex chordoma families at the NIH Clinical Center under protocol 78-C-0039. We also want to determine whether alterations in any identified chordoma susceptibility genes are associated with sporadic chordoma in the general population.

Objectives:

The major goal of this protocol is to identify sporadic chordoma patients willing to provide germline and tumor DNA for studies to determine the frequency of alterations in chordoma susceptibility genes. Our previous protocols with SEER and Massachusetts General Hospital to identify chordoma patients were limited to residents of specific geographic regions in the U.S. (2 states and 2 metropolitan areas) or to patients with pediatric skull base tumors. This protocol will enroll patients who more broadly represent the age, site and gender distributions of sporadic chordoma in the general U.S. population.

Eligibility:

Eligible patients are males and females in the U.S. with chordoma diagnosed at any age and at any primary site. Because we want to obtain saliva from all participants, eligibility is limited to patients who will be greater than or equal to age 6 years at the time of enrollment.

Design:

The study description and contacting information including an e-mail link to the study contact person will be posted on web sites of two chordoma support groups. We will mail study information to be given to patients to colleagues at major medical centers that treat chordoma.

The components of the study will be carried out in subjects' homes using materials mailed to them. Up to 100 participants will: 1) complete a self-administered Personal and Family Medical History Questionnaire, 2) collect saliva using a saliva collection kit, and 3) provide permission to obtain medical/pathology records, and paraffin blocks or slides on each primary chordoma. Parents will serve as proxies for minor children.

We will recontact patients who report chordoma in at least one blood relative. If we confirm the relative's chordoma diagnosis, we will invite the study subject and selected family members to participate in clinical and gene mapping studies under protocol 78-C-0039. We may also recontact study participants to tell them about any new studies on chordoma etiology. They can decide at that time whether they want to participate in them.

DETAILED DESCRIPTION:
Synopsis

Background: Chordoma is a rare, slow growing, often fatal bone cancer derived from remnants of the embryonic notochord. It occurs mostly in the axial skeleton (skull base, vertebrae, sacrum and coccyx), is more frequent in males than females, and has a median age at diagnosis of 58.5 years, with a wide age range. This typically sporadic tumor is often advanced at presentation, and mortality is high due to local recurrence or distant metastases. The usual treatment is surgery, followed by adjuvant radiation therapy. Chemotherapy has not had a significant treatment role.

Although most chordomas are sporadic, we previously identified germline duplication of the T gene (T-dup+), now designated TBXT, which encodes brachyury, a transcription factor that plays an important role in embryonic development, as a major susceptibility mechanism in familial chordoma. A common polymorphism in TBXT is also associated with an increased risk for both familial and sporadic chordoma. Although chordomas are slow-growing, local recurrences are common and treatment options are limited particularly for those with advanced disease. Thus, a better understanding of predisposing factors and molecular processes in chordoma is critically needed.

Objectives:

* To identify loci that cause susceptibility to chordoma and related tumors
* To determine the functional significance of mutations or other genetic changes at these loci
* To determine the frequency of alterations in chordoma susceptibility genes
* To identify genetic determinants conferring chordoma and related tumors risk in individuals
* To evaluate the natural history of disease in chordoma and related tumors, including evaluation of survival

Endpoints:

Primary Endpoint: All cancers that occur in individuals and families at high risk of chordoma

Secondary Endpoints: Markers of pre-malignant conditions such as benign notochordal cell tumors (BCNT), notochordal remnants

Study Population: Eligible patients are males and females in the U.S. or Canada with chordoma or related tumors diagnosed at any age and at any primary site. Because we want to obtain saliva from all participants, eligibility is limited to patients who will be > age 6 years at the time of enrolment.

Design of Sites/Facilities Enrolling Participants:

The components of the study will be carried out in subjects homes using materials mailed to them. The components include: 1) a self-administered Personal and Family Medical History Questionnaire, 2) saliva collected as a source of germline DNA using a saliva collection kit; 3) providing permission to obtain medical/pathology records, and paraffin blocks or slides on each primary ch ordoma and related tumors; 4) a self-administered Follow-Up Questionnaire to collect information about treatment, additional chordomas, and changes in health status since initial chordoma diagnosis.

Study Duration:

Start Date: 01/22/2011 End Date: 12/31/2051

This study is designed to be an open-ended natural history study with anticipated enrollment of 10-40 patients per year, with an accrual ceiling of 400.

Participant Duration:

Study participants may be reevaluated every few years to document changes in their history of chordoma over time and to collect information on treatment and survival. This is essential for establishing the natural history of chordoma and related tumors and to investigate the clinical significance of molecular subtypes.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:
* To be eligible subjects must be at least 6 years old at the time of enrollment, be the only person in their family ever diagnosed with chordoma, and reside in the U.S or Canada.
* Chordoma in the patients can have been diagnosed at any age and any primary site.

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible subjects include male and female patients diagnosed with Chordoma after 6 years of age. Participants may be located throughout the United States and Canada. The sample is a non-probability sample and eligible patients with Chordoma complete all study related activities by mail, after initial contact and determination of eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2011-01-02 (Actual)

PRIMARY OUTCOMES:
To determine the frequency of alterations in chordoma susceptibility genes in the general population | Multiple/ongoing
  - Susceptibility genes for Chordoma - Association between age at dx/Chordoma subtype and genetic risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Alisa M Goldstein, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Westat, Inc., Rockville, Maryland, United States

REFERENCES:
- [Background] Kelley MJ, Shi J, Ballew B, Hyland PL, Li WQ, Rotunno M, Alcorta DA, Liebsch NJ, Mitchell J, Bass S, Roberson D, Boland J, Cullen M, He J, Burdette L, Yeager M, Chanock SJ, Parry DM, Goldstein AM, Yang XR. Characterization of T gene sequence variants and germline duplications in familial and sporadic chordoma. Hum Genet. 2014 Oct;133(10):1289-97. doi: 10.1007/s00439-014-1463-z. Epub 2014 Jul 4. PMID 24990759
- [Background] Yang X', Beerman M, Bergen AW, Parry DM, Sheridan E, Liebsch NJ, Kelley MJ, Chanock S, Goldstein AM. Corroboration of a familial chordoma locus on chromosome 7q and evidence of genetic heterogeneity using single nucleotide polymorphisms (SNPs). Int J Cancer. 2005 Sep 1;116(3):487-91. doi: 10.1002/ijc.21006. PMID 15818627
- [Background] Yang XR, Ng D, Alcorta DA, Liebsch NJ, Sheridan E, Li S, Goldstein AM, Parry DM, Kelley MJ. T (brachyury) gene duplication confers major susceptibility to familial chordoma. Nat Genet. 2009 Nov;41(11):1176-8. doi: 10.1038/ng.454. Epub 2009 Oct 4. PMID 19801981